CLINICAL TRIAL: NCT01605942
Title: A Safety and Efficacy Study of a Dexamethasone Drug Delivery System for Postoperative Inflammation and Pain After Cataract Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to corporate decision.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 206207-027
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Results first posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone Drug Delivery System (Experimental): Dexamethasone Drug Delivery System administered into the study eye at the conclusion of cataract surgery on Day 1.
  Interventions: Drug: Dexamethasone Drug Delivery System
- Placebo Drug Delivery System (Placebo Comparator): Placebo Drug Delivery System administered into the study eye at the conclusion of cataract surgery on Day 1.
  Interventions: Drug: Placebo Drug Delivery System

INTERVENTIONS:
Drug: Dexamethasone Drug Delivery System — Dexamethasone Drug Delivery System administered into the study eye at the conclusion of cataract surgery on Day 1.
  Arms: Dexamethasone Drug Delivery System
Drug: Placebo Drug Delivery System — Placebo Drug Delivery System administered into the study eye at the conclusion of cataract surgery on Day 1.
  Arms: Placebo Drug Delivery System

SUMMARY:
This is a safety and efficacy study of a Dexamethasone Drug Delivery System for anterior segment inflammation and pain following cataract extraction with lens implantation.

ELIGIBILITY:
Inclusion Criteria:

* Planned single cataract extraction with lens implant
* Best-corrected visual acuity of 20/200 or better in the opposite eye

Exclusion Criteria:

* Glaucoma or history of intraocular hypertension in the study eye
* History of chronic ocular allergy in the last year requiring treatment
* Scheduled for cataract surgery in the non-study eye during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was terminated due to corporate decision and enrollment was not completed.
Period: Overall Study
Arm/Group | Dexamethasone Drug Delivery System | Placebo Drug Delivery System
Started | 6 | 2
Completed | 6 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone Drug Delivery System | Placebo Drug Delivery System | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Customized [Number; unit: Participants]
  <45 years | 0 | 0 | 0
  Between 45 and 65 years | 1 | 0 | 1
  >65 years | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clearance of Anterior Chamber Inflammation
Description: The anterior chamber is the area in front of the iris (colored part of the eye). Inflammation is measured on a scale ranging from 0 (best) to 8 (worst).
Time Frame: Up to Day 71
Population: Safety: all patients who received study treatment at randomization/surgery (day 1)
Measure: Number; unit: Patients
Arm/Group | Dexamethasone Drug Delivery System | Placebo Drug Delivery System
Number analyzed (Participants) | 6 | 2
Patients | 4 | 1

2. Secondary Outcome: Plasma Levels of Dexamethasone
Description: Levels of dexamethasone in plasma are evaluated. Plasma is the fluid portion of the blood.
Time Frame: Day 2, Day 7, Day 14
Population: Pharmacokinetic: all patients who received dexamethasone and consented to pharmacokinetic analysis.
Measure: Mean (Standard Deviation); unit: Nanograms/Milliliter (ng/mL)
Arm/Group | Dexamethasone Drug Delivery System
Number analyzed (Participants) | 6
Nanograms/Milliliter (ng/mL)
  Day 2 | 0.101 (0.038)
  Day 7 | 0 (NA) — Below the lower limit of quantitation
  Day 14 | 0 (NA) — Below the lower limit of quantitation

ADVERSE EVENTS:
Arm/Group | Dexamethasone Drug Delivery System | Placebo Drug Delivery System
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/2
Other Adverse Events (participants affected / at risk) | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone Drug Delivery System (N=6) | Placebo Drug Delivery System (N=2)
Corneal Oedema (Eye disorders) | 2 | 0
Retinal Tear (Eye disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone Drug Delivery System (N=6) | Placebo Drug Delivery System (N=2)
Anterior Chamber Cell (Eye disorders) | 6 | 2
Anterior Chamber Flare (Eye disorders) | 6 | 2
Corneal Oedema (Eye disorders) | 5 | 2
Conjunctival Oedema (Eye disorders) | 3 | 2
Corneal Deposits (Eye disorders) | 3 | 0
Intraocular Pressure Increased (Investigations) | 3 | 0
Iris Adhesions (Eye disorders) | 3 | 0
Punctate Keratitis (Eye disorders) | 3 | 0
Conjunctival Hyperaemia (Eye disorders) | 2 | 2
Visual Acuity Reduced (Eye disorders) | 2 | 1
Eye Pain (Eye disorders) | 2 | 0
Eye Pruritus (Eye disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Photophobia (Eye disorders) | 2 | 0
Facial Pain (General disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Conjunctival Haemorrhage (Eye disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Foreign Body Sensation in Eyes (Eye disorders) | 1 | 0
Glare (Eye disorders) | 1 | 0
Halo Vision (Eye disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Retinal Degeneration (Eye disorders) | 1 | 0
Retinal Tear (Eye disorders) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Vitreous Detachment (Eye disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Eyelid Oedema (Eye disorders) | 0 | 2
Eye Irritation (Eye disorders) | 0 | 1
Lacrimation Increased (Eye disorders) | 0 | 1
Photopsia (Eye disorders) | 0 | 1
Posterior Capsule Opacification (Eye disorders) | 0 | 1
Vitreous Floaters (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.